CLINICAL TRIAL: NCT01114581
Title: Evaluating the Effect of Mucinex 1200mg on Mucociliary and Cough Clearance During an Acute Respiratory Infection
Acronym: MCC/CC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-MUC-01
Record Dates: First submitted 2010-04-28; First posted 2010-05-03 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Acute Respiratory Infection
Keywords: Acute Respiratory Infection; Mucociliary; Cough Clearance; Guaifenesin
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Guaifenesin (Active Comparator): Mucinex 1200mg (Guaifenesin)given as 2, 600mg tablets
  Interventions: Drug: Mucinex
- Placebo (Placebo Comparator): Given as 2 tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mucinex — Mucinex 1200mg (Guaifenesin) given as 2,600mg tablets, one time on day 1 of the study
  Arms: Guaifenesin
Drug: Placebo — Placebo given as 2 tablets
  Arms: Placebo

SUMMARY:
The purpose of this research study is to explore the mechanism of action of Mucinex, an oral, over-the-counter, FDA approved expectorant in patients with acute respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of cough, thickened mucus and chest congestion
* Able to produce sputum
* Non Smoker

Exclusion Criteria:

* Pregnant
* Smokers
* Fever above 101°F
* Any chronic illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bennett, PhD, Principal Investigator — University of North Carolina
Locations (1):
- Center for Environmental Medicine, Asthma, and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Bennett WD, Kala A, Duckworth H, Zeman KL, Wu J, Henderson A, Yopp M, Rubin BK. Effect of a single 1200 Mg dose of Mucinex(R) on mucociliary and cough clearance during an acute respiratory tract infection. Respir Med. 2015 Nov;109(11):1476-83. doi: 10.1016/j.rmed.2015.09.017. Epub 2015 Oct 9. PMID 26462765

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Guaifenesin | Placebo
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guaifenesin | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (6.0) | 30.0 (11.94) | 27.9 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 10 | 9 | 19
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percent of Inhaled Radioactive Tracer Particles Cleared From Lungs
Description: Percentage of inhaled radioactive tracer (Ave180Clear)
Time Frame: 3 hours following inhalation of radioactive tracer particles
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: Percentage of inhaled radioactive tracer
Arm/Group | Guaifenesin | Placebo
Number analyzed (Participants) | 19 | 19
Percentage of inhaled radioactive tracer | 21.4 (99) | 23.1 (99)

2. Secondary Outcome: Guaifenesin AUC(0-3)
Time Frame: 3 hours following dose administration
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Guaifenesin | Placebo
Number analyzed (Participants) | 19 | 0
ng*hr/mL | 4060 (71) |

3. Secondary Outcome: Assess Sputum Properties (Objective Measures) and Symptoms (Subjective Measures) After Treatment With Mucinex or Placebo.
Time Frame: Within 10 days of developing symptoms associated with a respiratory tract infection
Population: The data for this secondary outcome cannot be reported as operational issues with the collection and transport of the samples occurred.
Arm/Group | Guaifenesin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Guaifenesin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less